CLINICAL TRIAL: NCT05222919
Title: Study to Evaluate the Efficacy of Bare Performance Nutrition's Peak Sleep Supplementation on Sleep Quality and Duration.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bare Performance Nutrition (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 20225
Record Dates: First submitted 2022-01-25; First posted 2022-02-03 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Sleep

STUDY DESIGN:
Intervention Model Description: single-blinded observational randomized-control trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bare performance supplement (Active Comparator): Dietary supplement
  Interventions: Dietary Supplement: Bare performance supplement
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Bare performance supplement — dietary supplement
  Arms: Bare performance supplement
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a single-blinded observational randomized-control trial to study the efficacy of a dietary supplement and its effect on sleep quality, recovery, and workout performance.

DETAILED DESCRIPTION:
This is a single-blinded observational randomized-control trial to study the efficacy of a dietary supplement and its effect on sleep quality, recovery, and workout performance.

It is hypothesized that the dietary supplement "Peak Sleep" will improve sleep quality - as defined as deep sleep, REM sleep, and feeling more rested the next day, as well as promoting the performance in workouts of trial participants.

A total of 72 participants will be recruited for the trial following the screening. The trial will be fully remote, a technology platform will be utilized to screen, enroll and capture study data of the participants, and participants will either receive the "Peak Sleep" product or receive a placebo - depending on the study group they got randomized in - for eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male & Female between 24-45 years old
* Self-reported mild to moderate sleep issues
* 3+ days of physical exercise per week
* Self-reported stressful lifestyle
* Own a sleep tracker that can be used for the study (e.g. Oura ring, Apple Watch, FitBit, -Whoop band, or similar other devices)
* Must be in good health (don't report any medical conditions asked in the screening questionnaire)
* Following a stable, consistent diet regimen
* Willing to maintain current dietary pattern, activity level, and stable body weight for the duration of the study, and refrain from any drastic lifestyle changes

Exclusion Criteria:

* Severe chronic conditions including oncological conditions, psychiatric disease, or other
* Diagnosed insomnia
* Food intolerances/allergies that require an EpiPen
* Females that are pregnant, want to become pregnant for the duration of the study, or who are breastfeeding
* Individuals that participate in another research study during the study period
* Individuals with a history of drug, alcohol, or substance abuse
* Individuals taking any other sleep supplements and are unwilling to stop taking those supplements for the duration of the study period
* Individuals who have night terrors regularly
* Individuals who regularly sleepwalk
* Individuals who have regular bad dreams

Ages: 24 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Change in sleep quality | Baseline to 8 weeks
  Survey-based assessment (0-5 scale with 0 being the lowest possible score and 5 being the highest) of changes in sleep quality between baseline and study intervention period.
Change in recovery time after a workout | Baseline to 8 weeks
  Survey-based assessment (0-5 scale with 0 being the lowest possible score and 5 being the highest) of changes in workout recovery time between baseline and study intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Mitschke, Principal Investigator — Citruslabs
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided